CLINICAL TRIAL: NCT02171000
Title: Safety, Pharmacokinetics and Pharmacodynamics After Multiple Oral Doses of BIBR 1048 MS Capsule (150 mg b.i.d., 7 Days) in Healthy Japanese Male Subjects (Open Label Study)
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics After Multiple Oral Doses of BIBR 1048 MS Capsule in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.55
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (1):
- BIBR 1048 (Experimental): BIBR 1048 MS
  Interventions: Drug: BIBR 1048 MS

INTERVENTIONS:
Drug: BIBR 1048 MS — 150 mg capsules, b.i.d, 7 days
  Other Names: dabigatran etexilate

SUMMARY:
To investigate safety, pharmacokinetics and pharmacodynamics of BIBR 1048 MS following oral administration of multiple doses (150 mg b.i.d., 7 days)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate and body temperature), 12-lead ECG, clinical laboratory tests
   * 1.1 No finding of clinical relevance
   * 1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥20 and Age ≤35 years
3. Body Mass Index (BMI) ≥18 and BMI <25 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the trial in accordance with Japanese GCP (Ministry of Health, Labour and Welfare Ordinance No.28, March 27, 1997).

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Subject was not able to use an adequate form of contraception from the time of the first dose on Day 1 up to end-of study examination
3. Diseases of the central nervous system (such as epilepsy), psychiatric disorders or neurological disorders
4. History of clinically significant orthostatic hypotension, clinically significant current or past fainting spells or blackouts.
5. Chronic or relevant acute infections
6. History of

   * allergy/hypersensitivity (including drug allergy) which was deemed relevant to the safety assessment as judged by the investigator (excluding asymptomatic seasonal rhinitis/hay fever)
   * any bleeding disorder including prolonged or habitual bleeding
   * other hematologic diseases
   * cerebral bleeding (e.g. after a car accident)
   * concussions (head trauma resulting in injuring to brain) with or without loss of consciousness
7. Intake of drugs with a long half-life (> 24 hours) within at least 1 month or less than 10 half-lives, whichever was shorter, of the respective drug prior to administration or during the trial
8. Use of aspirin (including over-the-counter medications), antiplatelet agents like ticlopidine or dipyridamole, chronic administration of non-steroidal anti-inflammatory drugs (NSAIDs, coumadin like anticoagulants, chronic use of corticosteroids, heparin or fibrinolytic agents within 14 days prior to administration up to end-of-study examination
9. Participation in another trial with an investigational drug within 3 months prior to administration up to end-of-study examination
10. Smoker (>10 cigarettes/day or inability to refrain from smoking during the trial)
11. Alcohol abuse (more than 60 g/day; confirmed by interview)
12. Drug abuse (confirmed by interview)
13. Blood donation (more than 100 mL from 3 months prior to screening and any blood donation from screening up to end-of-study examination)
14. Excessive physical activities (within 7 days prior to the first drug administration up to end-of-study examination)
15. Any laboratory value outside the reference range that was of clinical relevance
16. Known hypersensitivity to the investigational drug or its excipients
17. Subject who was judged ineligible by the investigator or the sub-investigator
18. History of any familial bleeding disorder
19. Thrombocytes < 15 x 104 /μL

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2005-04; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical examination | within 14 days prior to drug administration until up to 18 days post drug administration
Change from baseline in vital signs | within 14 days prior to drug administration until up to 18 days post drug administration
Change from baseline in 12-lead electrocardiogram (ECG) | within 14 days prior to drug administration until up to 18 days post drug administration
Change from baseline in clinical laboratory tests | within 14 days prior to drug administration until up to 18 days post drug administration
Number of participants with adverse events | within 14 days prior to drug administration until up to 18 days post drug administration

SECONDARY OUTCOMES:
Changes in activated partial thromboplastin time (aPTT) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Changes in ecarin clotting time (ECT) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Changes in thrombin time (TT) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Changes in prothrombin time expressed as international normalised ratio (INR) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Time from dosing to maximum measured concentration of the analyte in plasma (tmax) | Day 1 and 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 h after drug administration (morning), Day 2 to 6 prior drug administration (morning), Day 5 and 6 prior drug administration (evening), Day 7 24, 36, 48 h after final drug administration
Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the single dose on Day 1 (AUCτ,1) | Day 1 before, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours after drug administration in the morning
Amount of analyte that is eliminated in urine from the time point t1 to time point t2 ( Aet1-t2 ) | Day 1: 0-4, 4-8, 8-12 and 12-24 hours after the first drug administration, on Day 7: 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours after the last drug administration
Renal clearance of the analyte from the time point t1 until the time point t2 (CLR,t1-t2 ) | Day 1: 0-4, 4-8, 8-12 and 12-24 hours after the first drug administration, on Day 7: 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours after the last drug administration
Fraction of analyte eliminated in urine from time point t1 to time point t2 (fet1-t2) | Day 1: 0-4, 4-8, 8-12 and 12-24 hours after the first drug administration, on Day 7: 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours after the last drug administration
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Time from last dosing to maximum concentration of the analyte in plasma at steady state (tmax,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Terminal rate constant in plasma at steady state (λz,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Mean residence time of the analyte in the body at steady state after po administration (MRTpo,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration (CL/F,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Apparent volume of distribution during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration
Amount of analyte that is eliminated in urine at steady state from the time point t1 to time point t2 (Aet1-t2,ss) | Day 7 : 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours after the last drug administration
Fraction of analyte eliminated in urine at steady state from time point t1 to time point t2 (fet1-t2,ss) | Day 7: 0-4, 4-8, 8-12, 12-24, 24-48 and 48-72 hours after the last drug administration
Renal clearance of the analyte in plasma from the time point t1 until the time point t2 at steady state (CLR,t1-t2,ss) | Day 7 prior, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 hours after final drug administration